CLINICAL TRIAL: NCT01901263
Title: Initial and Long-term Evaluation of Patients With Behavioural Symptoms and Hospitalized in Cognitive and Behavioural Units
Brief Title: Patients With Behavioural Symptoms and Hospitalized in Cognitive and Behavioural Units
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Agence Régionale de Santé Rhône-Alpes (Other)
Responsible Party: Sponsor
Other Study IDs: 1208125; 13.069bis (Other: CCTIRS)
Record Dates: First submitted 2013-07-09; First posted 2013-07-17 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-07

CONDITIONS: Alzheimer Disease
Keywords: Cognitive and behavioral units; Alzheimer Disease; Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Amyloid beta-Protein Precursor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patient with alzheimer's disease: Cohort of patients with psychological symptoms of dementia hospitalised in Cognitive and Behaviorial Units (CBUs)
  Evaluation of these units through the observation of the behavioral and psychological symptoms of dementia evolution : NPI score, caregivers quality of life, caregivers burden, collection of psychotropic drugs, the rehospitalisation rate
  Interventions: Behavioral: patients with alzheimer's disease

INTERVENTIONS:
Behavioral: patients with alzheimer's disease — the Neuropsychiatric Inventory (NPI), is uded to assess 10 behavioral disturbances occurring in dementia patients: delusions, hallucinations, dysphoria, anxiety, agitation/aggression, euphoria, disinhibition, irritability/lability, apathy, and aberrant motor activity. The NPI uses a screening strategy to minimize administration time, examining and scoring only those behavioral domains with positive responses to screening questions.

SUMMARY:
Cognitive and behavioral units (CBUs) have been created between 2008 and 2012 French National Alzheimer plan for the management of behavior problems of patients suffering from Alzheimer's disease or other related disorders and necessitating hospitalisation. This Alzheimer plan is promoting the evaluation of these units through the observation of the behavioral and psychological symptoms of dementia (BPSD) evolution. As these units are new, it appears important to assess their long-term impact on patients care.

DETAILED DESCRIPTION:
EXPECTED RESULTS The present study should allow to better understand the long-term impact of CBU on care of patients with Alzheimer disease and BPSD. Moreover, it should allow to identify patients improved by CBU.

ELIGIBILITY:
Inclusion Criteria:

* patient hospitalized on CBUs
* patient with the diagnostic criteria for disease related to dementia stage with a Clinical Demential Rating ≥ 1
* patient with a caregiver who is fairly frequent contact with the patient in order to observe the appearance of behavior changes

Exclusion Criteria:

* Patient living alone at home
* Patient with risk of death within one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Alzheimer's disease or associated disorders and BDSP and hospitalized in a CBU
Sampling Method: Non-Probability Sample
Enrollment: 306 (Actual)
Dates: Start 2012-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Neuropsychiatric Inventory (NPI) score | one year
  impact of CBU effectiveness in reducing BPSD

SECONDARY OUTCOMES:
CBU effectiveness in reducing BPSD | 6 months
CBU effectiveness on quality of life of patients and caregivers, and on caregivers' burden | one year
Psychotropic drugs (in particular neuroleptic drugs) consumption | one year
rehospitalisation rate for BPSD of the patients in the year following their hospitalisation in CBU | one year

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle ROUCH, PhD, Principal Investigator — CHU de Saint-Etienne
Locations (3):
- France (3):
  - CH Saint Jean de Dieu, Lyon
  - CHU de Saint Etienne, Saint-Etienne
  - Hospices Civils de Lyon, Villeurbanne

REFERENCES:
- [Derived] Pongan E, Freulon M, Delphin-Combe F, Dibie-Racoupeau F, Martin-Gaujard G, Federico D, Waissi A, Richard G, Jacqueline S, Fabre F, Trombert-Paviot B, Krolak-Salmon P, Laurent B, Rouch I. Initial and long-term evaluation of patients with Alzheimer's after hospitalization in cognitive and behavioural units: the EVITAL study design. BMC Psychiatry. 2014 Nov 15;14:308. doi: 10.1186/s12888-014-0308-6. PMID 25398578